CLINICAL TRIAL: NCT04017377
Title: Study of Radiation Therapy With Concomitant Nab-paclitaxel and Cisplatin Chemotherapy in Patients With Locally Advanced Cervical Cancer
Brief Title: VMAT Concurrent Cisplatin Plus Nab-paclitaxel for Local Advanced Cervical Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Junjie Wang, Principal Investigator, Peking University Third Hospital
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M2019163
Record Dates: First submitted 2019-07-09; First posted 2019-07-12 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Cisplatin; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chemotherapy+ Radiation therapy (Experimental): Chemotherapy: Patients firstly receive an escalating dose of weekly Nab-paclitaxel starting at 10 mg/m^2 up to 70 mg/m^2, Patients secondly receive weekly cisplatin (40 mg/m^2). Treatment repeats every week until the disease recurrence or unacceptable toxicity, death or begin a novel therapeutic. Concurrent chemotherapy is a weekly regimen during radiotherapy. Patients will complete at least 4 cycles of concurrent chemoradiotherapy, until the maximal tolerated dose (MTD) appeared.
  Radiation therapy: Patients also receive pelvic radiation therapy once daily (Monday-Friday) for a total of 28 fractions and intracavitary brachytherapy twice a week for a total 5 fractions. Complete radiotherapy within 55 days.
  Interventions: Drug: Drug: Cisplatin; nab-paclitaxel

INTERVENTIONS:
Drug: Drug: Cisplatin; nab-paclitaxel — Drug: Paclitaxel for Injection（Albumin Bound). Other Name: Ke ai li, ZhusheyongZishanchun(Baidanbai Jiehexing)

SUMMARY:
This is a single arm, open-lable Phase I clinical trial. Eligible patients will have Histologically proven stage IB2-IVA cervical cancer. We hypothesize that Nab-paclitaxel in combination with cisplatin and radiotherapy may have anti-tumor activity in patients with cervical cancer. Nab-paclitaxel has not previously been combined with conventional RT-CT to treat cervical cancer.

DETAILED DESCRIPTION:
During the phase I study, patients will receive radiation therapy to pelvis (50.4 Gy in 28fractions), and followed by HDR intracavitary (30Gy in 5 fractions) brachytherapy. Concurrent chemotherapy was administered with weekly cisplatin (40 mg/m^2) and an escalating dose of weekly Nab-paclitaxel starting at 10 mg/m^2 up to 70 mg/m^2. Chemotherapy agents were administered in escalating doses to cohorts of three patients at each dose level.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years and ≤ 75 years.
* Patients with histologically confirmed newly diagnosed advanced cervical cancer (squamous cell carcinoma, adenocarcinoma, and adenosquamous cell carcinoma): Federation of Gynecology and Obstetrics (FIGO) clinical stages IB2-IVA.
* At least one measurable objective lesion was identified based on the RECIST1.1 criteria;
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2;
* The expected survival after surgery ≥ 3 months;
* LVEF≥55%;
* Bone marrow function: Neutrophils ≥ 1.5×10^9/L, platelets ≥ 100×10^9/L, and hemoglobin ≥ 90 g/L;
* Liver and renal function: Serum creatinine ≤ 1.5 times the upper limit of normal. AST and ALT ≤ 2.5 times the upper limit of normal Total bilirubin ≤ 1.5 times the upper limit of normal, or ≤ 2.5 times the upper limit of normal in patients with Gilbert's syndrome.
* Subjects of child-bearing age must agree to take effective contraceptive measures during the study period; Serum or urine pregnancy tests must be negative for women of childbearing age;
* Women must not lactate;
* Signed informed content obtained prior to treatment；

Exclusion Criteria:

* Patients previously treated with nab-paclitaxel;
* Patients previously undergoing abdominal or pelvic radiotherapy；
* Patients with CNS diseases or brain metastases；
* Other malignant tumors other than cervical cancer occurred in the past 5 years；
* Patients who had Grade 2 or above Peripheral neuropathy；
* Patients had uncontrolled serious medical condition that the investigator considered may affect the subject's to receive treatment under the study program, For example, patients with severe medical diseases, including severe heart disease, cerebrovascular disease, uncontrolled diabetes, uncontrolled hypertension, uncontrolled infection, active peptic ulcer, etc；
* Dementia, changing of mental state or any mental illness which could hinder understanding or informed consent or fill out questionnaires；
* History of allergy or hypersensitivity to any therapeutic ingredient；
* Combined with other malignant tumors excepted pancreatic cancer within the first 5 years of randomization, excepted well-treated basal cell or squamous cell carcinoma of the skin, localized prostate cancer after radical resection, and ductal carcinoma in situ of the breast after radical resection；
* Previously received systemic therapy for advanced/metastatic pancreatic cancer;
* Subjects who had previously been pathologically diagnosed with squamous cell carcinoma (no organ limitation) and received neoadjuvant/adjuvant therapy with taxa regimen；
* Patients who had Grade 2 or above Peripheral neuropathy；
* Known to be allergic, highly sensitive or intolerant to the study-related drugs or their excipients;
* Participation in any trial drug treatment or another interventional clinical trial 30 days before screening period；
* Severe infections including, but not limited to, complications of infection, bacteremia or severe pneumonia that require hospitalization within 4 weeks of study treatment initiation；
* Subjects had hepatitis b surface antigen (HBsAg)-positive and HBV- DNA titer in peripheral blood greater than or equal to 1000 copy number /L; If HBsAg is positive and the peripheral blood HBV-DNA <1000 copy number /L, the subjects will be eligible for inclusion if the investigator considers that chronic hepatitis b is stable and does not increase the risk of subjects；
* Human immunodeficiency virus (HIV)- or hepatitis C virus (HCV) positive patients；
* The researchers considered that there were other conditions that were not suitable for enrollment.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-06-15 (Estimated); Study Completion 2020-07-15 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose(MTD)/Recommended Dose(RD) | Up to 5 weeks
  Maximum Tolerated Dose (MTD) will be defined during the Dose Escalation Stage based on evaluation of the number of patients with Dose-limiting Toxicity (DLT). The MTD will be used to determine the Recommended Dose (RD).

SECONDARY OUTCOMES:
Number of patients with Dose Limiting Toxicity (DLT) | Up to 5 weeks
  Dose-limiting toxicity is defined as an adverse event that is considered to be drug-related and meets one of the Protocol definitions.
Objective response rate (ORR) | Up to 5 weeks
  ORR was assessed by the site Investigator using RECIST 1.1 and was defined as the percentage of patients with a confirmed overall response of CR or PR.

CONTACTS AND LOCATIONS:
Overall Officials: Junjie Wang, MD, PhD, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University 3rd Hospital, Beijing, Beijng, China

IPD SHARING:
Plan to Share IPD: No